CLINICAL TRIAL: NCT00721084
Title: Sleep, Energy Metabolism and Diabetes Risk
Brief Title: Fitness and Sleep in People With Family History of Type 2 Diabetes.
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16079A-S1; R01HL089637 (NIH)
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Sleep; Physical Fitness; Type 2 Diabetes
Keywords: short sleep duration; maximal aerobic capacity; body fat; visceral adiposity; activity-related energy expenditure; energy metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Reduced sleep: Habitual sleep duration of less than 6 hours per night on most days of the week and total sleep of less than 43 hours per week.
- Reference sleep: Habitual sleep duration between 7 and 8.5 hours per night on most days of the week and total sleep of at least 53 hours per week.

SUMMARY:
Currently, it is not known if the amount of nighttime sleep has any effect on the overall physical fitness, and on how much energy do people who have a relative with type 2 diabetes (parent, sibling, or grandparent) use to perform activities of daily living. This study will test the hypothesis that individual differences in nighttime sleep duration are related to differences in the amount of energy used to perform activities of daily living and the overall level of physical fitness of the individual.

DETAILED DESCRIPTION:
The study includes 2 weeks of monitoring of the participants' patterns of sleep and wakefulness at home. At the beginning of this period, all participants will undergo measurements of their body composition (lean tissue, bone and fat) and their metabolic rate at rest and after a standard meal. At that time, all participants will also drink a glass of water containing harmless non-radioactive dense forms of oxygen and hydrogen, small amounts of which are found in natural water. Several urine samples will be collected before and after the participants drink the water at the beginning of the study and again 14 days later in order to measure the amount of energy that was used by them during this time. Participants will also wear small wristwatch-like activity monitors on their wrist and around their waist as they follow their usual everyday activities and sleep-wake schedules at home. The recordings from these monitors combined with daily sleep logs will be used to determine when the participants slept and when they were awake. On the last day of the study, the participants will undergo MRI measurements of the distribution of fat in their abdomen and complete a graded exercise test on a treadmill or stationary bicycle in order to determine what is the most strenuous level of exercise that they can perform. A medical doctor will supervise all study procedures that are done in the research laboratory.

ELIGIBILITY:
Inclusion Criteria:

* regular sleep habits
* BMI 20 to 27 kg/m2
* at least one parent, sibling or grandparent with type 2 diabetes
* no regular exercise habits

Exclusion Criteria:

* active smoker
* night or shift work
* have highly variable sleep habits
* have a hormonal disorder
* have a sleep disorder
* have an active medical problem
* for women: use of birth control pills
* for women: irregular menstrual periods or pregnancy
* use of medications/compounds that can disrupt sleep

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy non-obese community-living men and women with a parent, sibling or grandparent who has type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Total energy expenditure | during a 2-week observation period

SECONDARY OUTCOMES:
Maximal aerobic capacity | at the end of the observation period
Amount and distribution of body fat | at the end of the observation period
Physical activity related energy expenditure | during a 2-week observation period

CONTACTS AND LOCATIONS:
Overall Officials: Plamen D Penev, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Darukhanavala A, Booth JN 3rd, Bromley L, Whitmore H, Imperial J, Penev PD. Changes in insulin secretion and action in adults with familial risk for type 2 diabetes who curtail their sleep. Diabetes Care. 2011 Oct;34(10):2259-64. doi: 10.2337/dc11-0777. Epub 2011 Aug 11. PMID 21836106